CLINICAL TRIAL: NCT00837941
Title: Qualification of Single Dose Administration of Analgesic Therapy in the Treatment of Chronic Neuropathic Pain in Patients With Painful Diabetic Neuropathy
Brief Title: A Study of Single Dose Pain Therapy in Patients With Painful Diabetic Neuropathy (0000-115)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-115; 2009_515
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Painful Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): sequence 1 - Pregabalin, Duloxetine hydrochloride, Diphenhydramine hydrochloride
  Interventions: Drug: Comparator: A: Pregabalin; Drug: Comparator: B: Duloxetine; Drug: Comparator: C: Diphenhydramine hydrochloride
- 2 (Experimental): sequence 2 - Duloxetine hydrochloride, Pregabalin, Diphenhydramine hydrochloride
  Interventions: Drug: Comparator: A: Pregabalin; Drug: Comparator: B: Duloxetine; Drug: Comparator: C: Diphenhydramine hydrochloride
- 3 (Experimental): sequence 3 - Diphenhydramine hydrochloride, Duloxetine hydrochloride, Pregabalin
  Interventions: Drug: Comparator: A: Pregabalin; Drug: Comparator: B: Duloxetine; Drug: Comparator: C: Diphenhydramine hydrochloride
- 4 (Experimental): sequence 4 - Pregabalin, Diphenhydramine hydrochloride, Duloxetine hydrochloride
  Interventions: Drug: Comparator: A: Pregabalin; Drug: Comparator: B: Duloxetine; Drug: Comparator: C: Diphenhydramine hydrochloride
- 5 (Experimental): sequence 5 - Duloxetine hydrochloride, Diphenhydramine hydrochloride, Pregabalin
  Interventions: Drug: Comparator: A: Pregabalin; Drug: Comparator: B: Duloxetine; Drug: Comparator: C: Diphenhydramine hydrochloride
- 6 (Experimental): sequence 6 - Diphenhydramine hydrochloride, Pregabalin, Duloxetine hydrochloride
  Interventions: Drug: Comparator: A: Pregabalin; Drug: Comparator: B: Duloxetine; Drug: Comparator: C: Diphenhydramine hydrochloride

INTERVENTIONS:
Drug: Comparator: A: Pregabalin — 1 Pregabalin 300 mg capsule
Drug: Comparator: B: Duloxetine — 1 Duloxetine hydrochloride 60 mg capsule
Drug: Comparator: C: Diphenhydramine hydrochloride — 1 Diphenhydramine hydrochloride 25mg capsule

SUMMARY:
The purpose of this study is to determine if analgesic efficacy can be detected with single dose administration in patients with chronic neuropathic pain due to painful diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been treated for type 1 or 2 diabetes mellitus with glycosylated hemoglobin
* Patient has pain in both feet that occurred after onset of diabetes
* Patient agrees to maintain a consistent activity level throughout the study
* Patient is not on chronic pain therapy, or is on a stable dose of one pain therapy
* Female patients of reproductive potential must agree to use two acceptable methods of birth control through out the study
* Patients taking a pain medication must be on a stable dose at least 1 month prior to participating in study

Exclusion Criteria:

* Patient has a history of congestive heart failure
* Patient has/had a seizure disorder
* Patient has tried and failed 3 or more drugs to treat neuropathic pain
* Patient is currently taking pregabalin or duloxetine hydrochloride
* Patient has had a malignancy within the past 2 years (excluding basal cell carcinoma)
* Patient has history of hepatitis B or C or HIV infection
* Patient has skin-condition that may decrease sensitivity in area of neuropathic pain

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
analgesic efficacy measured by patients self reported pain level after single dose administration | 5-11 hours after single dose is administered

SECONDARY OUTCOMES:
The onset of analgesic efficacy following single dose of pregabalin and duloxetine hydrochloride versus placebo | 24 hours after single dose is administered

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC